CLINICAL TRIAL: NCT04245553
Title: Does Point of Care Ultrasound Change Needle Insertion Location During Routine Bedside Paracentesis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven Montague (Other)
Responsible Party: Sponsor-Investigator, Steven Montague, Medical Doctor, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 6028481
Record Dates: First submitted 2020-01-25; First posted 2020-01-29 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Ascites; Paracentesis; Point of Care Ultrasound (POCUS)
Keywords: Paracentesis; Point of Care Ultrasound (POCUS)
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental)
  Interventions: Diagnostic Test: Abdominal Point of Care Ultrasound

INTERVENTIONS:
Diagnostic Test: Abdominal Point of Care Ultrasound — Participants will be have their needle insertion site for a paracentesis land-marked using both the traditional anatomical method, and with a point of care ultrasound. Note that the current standard of care does not require the use of point of care ultrasound.

SUMMARY:
Paracentesis is a bedside procedure in which a needle is inserted into a patient's peritoneum in order to obtain ascitic fluid. This is a safe bedside procedure with very low risks of complications that is usually performed using physical exam maneuvers to determine the site of needle insertion. Point of care ultrasound (POCUS) technology has improved the safety of central venous catheter insertion and thoracentesis, yet the data on safety in paracentesis is equivocal. In a practical study, we aim to determine if POCUS will change the needle insertion site over the traditional anatomic landmarking method. Operators will landmark for paracentesis using conventional physical exam and then utilize POCUS to determine if there is a more optimal site. The primary endpoint will be whether POCUS yielded a change in the needle insertion site, as defined by a location greater than 5cm from the anatomic site, at least 20% of the time. The results will further our understanding of POCUS in improving procedural safety, thereby adding to the currently limited literature on this topic. Furthermore, this study will inform residency training programs about the utility in POCUS training for paracentesis and may advocate for the availability of POCUS devices to physicians performing this procedure.

ELIGIBILITY:
This is in effort to capture routine paracentesis cases.

Inclusion Criteria:

* Participants scheduled to have either a diagnostic of therapeutic paracentesis.
* Participants can be either inpatients under the care of general internal medicine, or outpatients under the care of gastroenterology or general internal medicine.
* Operators will be recruited on a volunteer basis and will include medical residents or subspecialty fellows with knowledge of POCUS for paracentesis purposes, either through core residency programs or more advanced training.

Exclusion Criteria:

* Loculated ascites
* Current anticoagulation
* Hemodynamic instability
* Bowel obstruction
* Pregnancy
* Abdominal wall cellulitis
* Platelet count <20

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Preference of land-marking method | Determined immediatly after the POCUS landmarking is done.
  Does the clinician performing the procedure prefer the needle insertion site found using point of care ultrasound, or using the traditional anatomic method. A clinically significant difference in location is defined as greater than or equal to 5cm apart. If the difference in locations is not at least 5cm apart, this will be defined as no preference in land-marking methods.

SECONDARY OUTCOMES:
Depth of Ascitis | Determined immediatly after the POCUS landmarking is done.
  Depth of ascitis, measured perpendicular to the overlying skin, at the location land-marked using traditional anatomic method, versus the location found with point of care ultrasound.
Immediate Complications | Occuring at any time between the needle insertion and removal of the paracentesis drain.
  The overall rate of any complications observed while performing the procedure. This includes bleeding, perforation/puncture of any internal organ, or a failed attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Montague, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Center, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No